CLINICAL TRIAL: NCT00723086
Title: An Extension Multicenter Phase II Open Label Non-comparative Trial of RP56976 Administered Every Three Weeks in Combination With Daily Prednisolone for Metastatic Hormone Refractory Prostate Cancer.
Brief Title: Japanese Study of the Combined Administration of Docetaxel With Prednisolone for Metastatic Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD6563; XRP6976J/2102
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Therapy, Prostatic Neoplasms
Keywords: docetaxel, prednisolone, drug combination
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel (XRP6976) — combined treatment with prednisolone

SUMMARY:
The purpose of this study is to evaluate the safety of docetaxel administered every 3 weeks repeatedly for 11 and more cycles and in combination with daily prednisolone for metastatic hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients who completed the 10 cycles of docetaxel administrations in the preceding XRP6976J/2101 study and wish to continue docetaxel administrations,and who have no alternative therapy for hormone refractory prostate cancer according to the Investigator's judgment.

Exclusion Criteria:

* Continuation in the study would be detrimental to the patient's well-being
* Development of life-threatening and/or toxic conditions not manageable by symptomatic care, dose reduction, or delay of dosing
* Obvious disease progression (rising prostate specific antigen, any increase of ≥ 20 % in the sum of the measurable lesion in comparison to the nadir value, and progression in non-measurable lesion)
* Patients treated with anti-cancer treatment other than study therapy after completion of 10 cycles of study treatment in the XRP6976J/2101 study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events on each grade evaluated by National Cancer Institute Common Toxicity Criteria (Version 2.0) | First treatment up to 37 months

SECONDARY OUTCOMES:
No obvious disease progression | First treatment up to 37 months

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan